CLINICAL TRIAL: NCT02527317
Title: An Observational Study of Dose Dense Chemotherapy With Lipegfilgrastim Support
Brief Title: Dose Dense Chemotherapy With Lipegfilgrastim Support in Early Breast Cancer
Status: Completed | Type: Observational
Sponsor: Beaumont Hospital (Other)
Responsible Party: Principal Investigator, Patrick Morris, Consultant Medical Oncologist, Beaumont Hospital
Other Study IDs: B1010
Record Dates: First submitted 2015-06-03; First posted 2015-08-19 (Estimated); Last update posted 2018-02-09 (Actual); Status verified 2018-02

CONDITIONS: Breast Cancer
Keywords: Early
MeSH Terms: conditions — Breast Neoplasms | interventions — pegfilgrastim

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Lipegfilgrastim — Investigate the incidence of treatment-related neutropenia following four cycles of dose dense (every 2 week) doxorubicin cyclophosphamide (AC) with lipegfilgrastim support (8 weeks).
  Other Names: Lonquex

SUMMARY:
This is a prospective, non-interventional, single arm study, which is examining doxorubicin and cyclophosphamide (AC) once every 2 weeks with lipegfilgrastim support in early breast cancer.

DETAILED DESCRIPTION:
An important advance in the use of dose dense chemotherapy regimens for breast cancer was the development of pegylated form of G-CSF (pegfilgrastim and lipegfilgrastim), which offered the convenience of single subcutaneous injection, rather than multiple daily injections

Lipegfilgrastim is a pegylated long-acting covalent conjugate of filgrastim (G-CSF). In a pivotal randomized phase III study in breast cancer lipegfilgrastim was shown to be non-inferior to pegfilgrastim.

In this prospective observational study the incidence of treatment-related neutropenia following four cycles of dose dense (every 2 week) doxorubicin cyclophosphamide (AC) with lipegfilgrastim support is being investigated.

Data will be collected on 40 consecutive patients treated with AC and lipegfilgrastim in Ireland.

The primary objective of this study is to determine the incidence of treatment-related neutropenia following four cycles of dose dense doxorubicin cyclophosphamide (AC) with lipegfilgrastim support (8 weeks).

Secondary Objectives

1. Determine the incidence of febrile neutropenia during 4 cycles (8 weeks)of dose dense AC with lipegfilgrastim
2. Examine the incidence of treatment-related neutropenia during subsequent intravenous cancer therapy up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Stage I-III Breast Cancer
3. Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1(see below)
4. Adequate Bone Marrow Function as defined by neutrophil count of ≥1.0 and platelet count of ≥ 100
5. Planned chemotherapy with Dose Dense Doxorubicin-Cyclophosphamide (AC) as deemed appropriate by a Consultant Medical Oncologist

General Indications for Dose Dense AC include:

1. T3 or T4 Tumours
2. N1 - N3 (Node Positive) Disease
3. Human Epidermal Growth Factor Receptor 2 (HER2) Positive Tumours.
4. Triple Negative Breast Cancer as evidenced by lack of expression of the estrogen receptor (ER), progesterone receptor (PR) and HER2

Exclusion Criteria:

1. Stage IV Breast Cancer
2. Pregnancy
3. Previous Chemotherapy Exposure
4. Prior Exposure to G-CSF
5. Known positive HIV Status
6. Cardiac or other concurrent illness, which at the investigator's discretion contraindicates the use of AC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Planned chemotherapy with Dose Dense Doxorubicin-Cyclophosphamide (AC) for early breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
incidence of treatment-related neutropenia | four cycles of dose dense doxorubicin cyclophosphamide (AC) with lipegfilgrastim support (8 weeks).
  The primary objective of this study is to determine the incidence of treatment-related neutropenia following four cycles of dose dense doxorubicin cyclophosphamide (AC) with lipegfilgrastim support (8 weeks).

SECONDARY OUTCOMES:
incidence of febrile neutropenia | four cycles of dose dense doxorubicin cyclophosphamide (AC) with lipegfilgrastim support (8 weeks).
  Determine the incidence of febrile neutropenia during 4 cycles (8 weeks) of dose dense AC with lipegfilgrastim
incidence of treatment-related neutropenia | Up to 1 year of subsequent chemotherapy
  Determine the incidence of treatment-related neutropenia during subsequent chemotherapy (up to 1 year)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick G Patrick, MD, Principal Investigator — Beaumont Hospital
Locations (1):
- Beaumont Hospital, Dublin, Ireland